CLINICAL TRIAL: NCT05438862
Title: Early Aortic Valve Surgery Versus Watchful Waiting Strategy in Severe Asymptomatic Aortic Regurgitation
Acronym: ELEANOR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Na Homolce Hospital (Other)
Collaborators: University Hospital Hradec Kralove (Other); Centre of Cardiovascular and Transplantation Surgery, Czech Republic (Other); St. Anne's University Hospital Brno, Czech Republic (Other); VZW Cardiovascular Research Center Aalst (Other); General University Hospital, Prague (Other); University Clinical Centre of Republic of Srpska (Other); AGEL Třinec-Podlesí Hospital (Unknown)
Responsible Party: Principal Investigator, Radka Kockova, MD, Ph.D., Associate Professor, Na Homolce Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6.4.2022/5
Record Dates: First submitted 2022-06-21; First posted 2022-06-30 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Aortic Valve Regurgitation
Keywords: aortic regurgitation; cardiac magnetic resonance; echocardiography; early surgical intervention
MeSH Terms: conditions — Aortic Valve Insufficiency

STUDY DESIGN:
Intervention Model Description: Randomization between early surgical and conventional watchful waiting strategy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early surgery (Experimental): Early surgical treatment, state of art aortic valve surgery.
  Interventions: Procedure: State of art aortic valve surgery
- Watchful waiting (No Intervention): Watchful waiting strategy, regular follow-up of patients with severe valve disease. Guideline-based indication for surgery only during the follow-up.

INTERVENTIONS:
Procedure: State of art aortic valve surgery — Optimal surgical treatment (aortic valve-sparing surgery, aortic valve replacement, Ross procedure).
  Arms: Early surgery

SUMMARY:
The optimal timing of surgical intervention in asymptomatic patients with severe aortic regurgitation remains controversial. As per cardiac magnetic resonance assessment, early surgical treatment will be compared with conventional guideline-based strategy in asymptomatic patients with severe aortic regurgitation.

DETAILED DESCRIPTION:
Introduction:

Aortic regurgitation (AR) is the third most frequent valvular heart disease in Western countries affecting rather young patients, mostly men. The degenerative process on the trileaflet aortic valve is the main cause of AR, followed by a congenital valve disease, typically bicuspid aortic valve. The high prevalence of bicuspid aortic valve in the general population which is frequently associated with aortic dilatation, another important cause of AR, can explain the unusual distribution of significant AR mainly among the population of males in their average 5th decade. Infective or rheumatic endocarditis and aortic dissection are less frequent reasons for AR.

Hemodynamically significant AR leads to volume and pressure overload of the left ventricle (LV). Severe LV dilatation and moderate LV hypertrophy are the main compensatory mechanisms that help to maintain cardiac output and relieve the increased LV wall stress. Doubling the cardiomyocyte size is accompanied by an increase in extracellular volume, including multiplying collagen fibres and increasing the volume of the non-collagen extracellular matrix. Untreated severe AR leads to advanced LV remodeling and LV dysfunction causing the development of heart failure.

The only appropriate treatment for chronic haemodynamically significant AR is aortic valve surgery. The indications for AR surgical treatment are summarized in the 2021 ESC/EATS Guidelines for the management of the valvular disease. Class I indications of aortic valve surgery are based on the presence of symptoms of heart failure (exertional dyspnoea, chest tightness) and/or presence of severe LV remodelling (LV ejection fraction ≤50% or LV end-systolic diameter (ESD) >50 mm or LV ESD Index >25 mm/m2 in patients with small body size). There is increasing evidence that patients undergoing surgery at such an advanced stage of the disease have already irreversible myocardial damage. There is also evidence that surgical risk in a relatively younger and low-risk population has decreased with novel surgical techniques and perioperative care, including aortic valve-sparing surgery with documented excellent long-term effects. Concerning these facts, it might be reasonable to shift the surgical treatment towards an earlier stage of the disease.

Available evidence including our study suggests higher clinical accuracy of cardiac magnetic resonance (CMR)-derived AR quantification than that of the guidelines-based echocardiographic (ECHO) Integrative approach (12-14). Severe AR defined as regurgitation fraction (RF) >33% and/or regurgitant volume (RV) >44 ml with LV dilatation defined as LV end-diastolic volume index (LVEDVI) >123 ml/m2 present the most accurate marker of early disease progression requiring surgery in a median of 399 (IQR 209) days (unpublished data).

Project Hypothesis:

1. We hypothesize that early surgical treatment will lead to early LV reverse remodeling, leading to the complete normalization of LV structure and function.
2. We hypothesize that early surgical treatment in patients with low surgical risk and severe AR as per CMR assessment will be a superior, safe procedure with a low incidence of early and late periprocedural complications in comparison to standard published data from large centres.
3. We hypothesize that early surgical treatment will lead to early improvement in quality of life and exercise performance in the majority of patients.
4. We hypothesize that early surgical treatment will be associated with lower long-term cardiovascular morbidity.

Project Plan:

1. All consecutive patients referred to the participating centre for a hemodynamically significant chronic AR will be screened. Patients with AR grade 3 and grade 4 without an indication for aortic valve surgery as per current Guidelines and who comply with the inclusion and exclusion criteria will be offered to participate in the study.
2. All patients will undergo CMR at baseline and after 12 months, including T1 mapping, contrast-enhanced imaging and flow sequence measurement at sinotubular junction according to study protocol in a particular centre. All CMR studies will be anonymized and digitally transferred to CoreLab based in University Hospital Hradec Králové. The off-line analysis will consist of the left and right ventricular volumes, mass and ejection fraction calculation. AR will be quantified utilising flow sequence measurement at the sinotubular junction. A correction for Eddy's current will be applied. Native T1 relaxation time will be measured in the midventricular septum.
3. All patients will undergo a comprehensive 2-dimensional (2D) and 3-dimensional (3D) ECHO at baseline and every six months of follow-up in each participating centre. Echocardiography will be performed using Vivid 7, Vivid E9, and Vivid E95 (GE Healthcare, Horten, Norway) to allow for advanced analysis. The off-line analysis will include the left ventricular volume, mass, ejection fraction and global longitudinal strain calculation. Aortic regurgitation will be quantified utilizing a widely accepted Integrative approach. Vena contracta area will be measured whenever possible. Moreover, baseline and 12-month images will be analysed centrally by one operator (Cardiovascular Center, Aalst, Belgium).
4. All patients will undergo 12-lead electrocardiography (ECG) and blood sample analysis at baseline and every six months of follow-up in each participating centre. One blood sample (serum and plasma) will be stored frozen at -80 C° for further analysis.
5. All patients will undergo an exercise stress test - spiroergometry (CPET) - at baseline and a 12-month follow-up in each participating centre. CPET will be used to validate asymptomatic status and to assess changes in exercise performance during follow-up.
6. All patients will fill out the questionnaire (RAND 36-Item Health Survey 1.0 Questionnaire Items) at baseline and 12 months after randomization.

6. Randomization will be computer-based, utilizing the covariate adaptive randomization method to achieve a balanced distribution of both patients' groups in between participating centres, age and gender.

7. Aortic valve surgery will be performed in each participating centre by an experienced surgeon who is a member of the study team. The type of surgery will be based on a "state of art" approach and local expertise with the preference for valve-sparing surgery or Ross procedure in carefully selected patients. Transesophageal ECHO will be performed in all patients to evaluate valve morphology and suitability for valve-sparing surgery. The surgery will be scheduled within 3 months after randomization for early surgery. Patients in the watchful waiting group study arm will undergo surgical treatment in agreement with current Guidelines for the disease progression during the study follow-up.

Methods:

Design The study will be prospective, randomized and multicenter, including international collaboration. Imaging data will be analyzed in a CoreLab based in the Czech Republic for CMR data (Faculty Hospital Hradec Králové) and Belgium for ECHO data (Cardiovascular Center Aalst).

Patients Patients with chronic grade 3 and grade 4 AR without an indication for surgical treatment as per current Guidelines will be enrolled in the study after signing the informed consent. The baseline examination consists of a clinical examination, ECG, blood test analysis (including N-terminal pro-brain natriuretic peptide), a comprehensive 2D and 3D ECHO, exercise stress test (CPET preferably) and CMR.

Patients with CMR-derived RF >35% or RV >45 ml and LV EDVI >125 mL/m2 will be randomised in a 1:1 ratio between early surgery (Group A) or watchful waiting (Group B). Patients, not fulfilling these CMR criteria, will enter the registry (Group C).

Patients in Group A will undergo aortic valve surgery within 3 months after randomisation. Their follow-up will consist of a repeat CMR and spiroergometry 12 months after enrolment. The regular follow-up will be every 6 months including a clinical examination, 2D and 3D ECHO and blood tests. Patients who will decline early surgical treatment might be reassigned to Group B but the total number must not exceed 6% of the total number of enrolled patients in a particular centre. The results will be statistically tested for both, intention to treat and as treated.

Patients in Group B and C will be reviewed every 6 months including a clinical examination, 2D and 3D ECHO and blood tests. A repeat CMR study and spiroergometry will be performed 12 months after enrolment. Patients who develop an indication for aortic valve surgery as per current Guidelines during the watchful waiting period of the study will undergo aortic valve surgery within 3 months after the onset of the indication.

ELIGIBILITY:
Inclusion Criteria:

* Chronic asymptomatic aortic regurgitation grade 3 (moderate to severe) and grade 4 (severe)
* No indication for the surgical treatment at the time of enrolment
* LV ejection fraction >50%
* Absence of more than mild-to-moderate concomitant valve disease or complex congenital heart disease

Exclusion Criteria:

* Age <18 years
* Clearance Creatinine <30 mL/min
* Contraindication for magnetic resonance (implanted active device, ferromagnetic implant incompatible with magnetic resonance scanner, cerebral aneurysm clip, metallic fragment in the eye or near sensitive tissue)
* Pregnancy
* Permanent atrial fibrillation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 217 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Composite safety and efficacy endpoint at 12 months post-randomization (all 3 criteria must be fulfilled): | 12 months
  1. Reverse LV remodelling (CMR-derived EDVI decrease >15% compared to baseline)
  2. LV ejection fraction >50%
  3. Absence of MACE (cardiovascular mortality, stroke, myocardial infarction, heart failure, infective endocarditis)

SECONDARY OUTCOMES:
Change in comparison to baseline: | 12 months
  1) Quality of life questionnaire >10%
Change in comparison to baseline: | 12 months
  2) Spiroergometry - maximal oxygen consumption (VO2 max) >10% and/or >3 ml/kg/min
Normalization of N-terminal pro B-natriuretic peptide serum level | 12 months
  NT-proBNP <112 ng/L
In hospital and 30 days mortality | 30 day postoperatively
  Perioperative and/or early postoperative mortality
Time to cardiovascular death | 12 months
  Death due to myocardial infarction, death due to heart failure, death due to stroke, death due to CV procedures, death due to CV hemorrhage, and sudden cardiac death.
Time to first heart failure hospitalization | 12 months
  Heart failure symptoms that require hospitalization.
Number of Participants with Major bleeding | 12 months
  Fatal bleeding, and/or symptomatic bleeding in a critical area or organ, such as intracranial, intraspinal, intraocular, retroperitoneal, intra-articular or pericardial, or intramuscular with compartment syndrome, and/or bleeding leading to transfusion of two or more units of whole blood or red cells.

CONTACTS AND LOCATIONS:
Overall Officials: Radka Kočková, MD, PhD, Principal Investigator — Na Homolce Hospital; Jan Vojáček, MD, PhD, Principal Investigator — Faculty Hospital Hradec Králové; Martin Pěnička, MD, PhD, Principal Investigator — Cardiovascular Center OLV Clinic
Locations (8):
- Cardiovascular Center OLV Clinic Aalst, Aalst, Belgium
- Czechia (6):
  - International Clinical Research Center, St. Anne´s University Hospital Brno, Brno
  - Center of Cardiovascular and Transplant Surgery, Brno
  - University Hospital Hradec Králové, Hradec Králové
  - 2nd Department of Internal Cardiovascular Medicine, First Faculty of Medicine, Charles University and General University Hospital in Prague, Prague
  - Na Homolce Hospital, Prague
  - Nemocnice AGEL Třinec-Podlesí, Třinec
- University Clinical Center of Serbia, Belgrade, Serbia

IPD SHARING:
Plan to Share IPD: Yes
Publication of the rationale and design of the study.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 12 months
Access Criteria: National Library of Medicine
URL: http://pubmed.ncbi.nlm.nih.gov/

REFERENCES:
- [Result] Iung B, Delgado V, Rosenhek R, Price S, Prendergast B, Wendler O, De Bonis M, Tribouilloy C, Evangelista A, Bogachev-Prokophiev A, Apor A, Ince H, Laroche C, Popescu BA, Pierard L, Haude M, Hindricks G, Ruschitzka F, Windecker S, Bax JJ, Maggioni A, Vahanian A; EORP VHD II Investigators. Contemporary Presentation and Management of Valvular Heart Disease: The EURObservational Research Programme Valvular Heart Disease II Survey. Circulation. 2019 Oct;140(14):1156-1169. doi: 10.1161/CIRCULATIONAHA.119.041080. Epub 2019 Sep 12. PMID 31510787
- [Result] Vahanian A, Beyersdorf F, Praz F, Milojevic M, Baldus S, Bauersachs J, Capodanno D, Conradi L, De Bonis M, De Paulis R, Delgado V, Freemantle N, Gilard M, Haugaa KH, Jeppsson A, Juni P, Pierard L, Prendergast BD, Sadaba JR, Tribouilloy C, Wojakowski W; ESC/EACTS Scientific Document Group. 2021 ESC/EACTS Guidelines for the management of valvular heart disease. Eur Heart J. 2022 Feb 12;43(7):561-632. doi: 10.1093/eurheartj/ehab395. No abstract available. PMID 34453165
- [Result] Michelena HI, Prakash SK, Della Corte A, Bissell MM, Anavekar N, Mathieu P, Bosse Y, Limongelli G, Bossone E, Benson DW, Lancellotti P, Isselbacher EM, Enriquez-Sarano M, Sundt TM 3rd, Pibarot P, Evangelista A, Milewicz DM, Body SC; BAVCon Investigators. Bicuspid aortic valve: identifying knowledge gaps and rising to the challenge from the International Bicuspid Aortic Valve Consortium (BAVCon). Circulation. 2014 Jun 24;129(25):2691-704. doi: 10.1161/CIRCULATIONAHA.113.007851. No abstract available. PMID 24958752
- [Result] Carabello BA. The relationship of left ventricular geometry and hypertrophy to left ventricular function in valvular heart disease. J Heart Valve Dis. 1995 Oct;4 Suppl 2:S132-8; discussion S138-9. PMID 8563989
- [Result] Villari B, Campbell SE, Hess OM, Mall G, Vassalli G, Weber KT, Krayenbuehl HP. Influence of collagen network on left ventricular systolic and diastolic function in aortic valve disease. J Am Coll Cardiol. 1993 Nov 1;22(5):1477-84. doi: 10.1016/0735-1097(93)90560-n. PMID 8227808
- [Result] de Meester C, Gerber BL, Vancraeynest D, Pouleur AC, Noirhomme P, Pasquet A, de Kerchove L, El Khoury G, Vanoverschelde JL. Do Guideline-Based Indications Result in an Outcome Penalty for Patients With Severe Aortic Regurgitation? JACC Cardiovasc Imaging. 2019 Nov;12(11 Pt 1):2126-2138. doi: 10.1016/j.jcmg.2018.11.022. Epub 2019 Jan 16. PMID 30660551
- [Result] Desai MY. Aortic regurgitation: are we operating too late? Ann Cardiothorac Surg. 2019 May;8(3):390-392. doi: 10.21037/acs.2019.04.06. No abstract available. PMID 31240183
- [Result] Dujardin KS, Enriquez-Sarano M, Schaff HV, Bailey KR, Seward JB, Tajik AJ. Mortality and morbidity of aortic regurgitation in clinical practice. A long-term follow-up study. Circulation. 1999 Apr 13;99(14):1851-7. doi: 10.1161/01.cir.99.14.1851. PMID 10199882
- [Result] Mentias A, Feng K, Alashi A, Rodriguez LL, Gillinov AM, Johnston DR, Sabik JF, Svensson LG, Grimm RA, Griffin BP, Desai MY. Long-Term Outcomes in Patients With Aortic Regurgitation and Preserved Left Ventricular Ejection Fraction. J Am Coll Cardiol. 2016 Nov 15;68(20):2144-2153. doi: 10.1016/j.jacc.2016.08.045. PMID 27855803
- [Result] David TE, Feindel CM, Webb GD, Colman JM, Armstrong S, Maganti M. Long-term results of aortic valve-sparing operations for aortic root aneurysm. J Thorac Cardiovasc Surg. 2006 Aug;132(2):347-54. doi: 10.1016/j.jtcvs.2006.03.053. Epub 2006 Jul 10. PMID 16872961
- [Result] Lansac E, de Kerchove L. Aortic valve repair techniques: state of the art. Eur J Cardiothorac Surg. 2018 Jun 1;53(6):1101-1107. doi: 10.1093/ejcts/ezy176. No abstract available. PMID 29718164
- [Result] Myerson SG, d'Arcy J, Mohiaddin R, Greenwood JP, Karamitsos TD, Francis JM, Banning AP, Christiansen JP, Neubauer S. Aortic regurgitation quantification using cardiovascular magnetic resonance: association with clinical outcome. Circulation. 2012 Sep 18;126(12):1452-60. doi: 10.1161/CIRCULATIONAHA.111.083600. Epub 2012 Aug 9. PMID 22879371
- [Result] Kockova R, Linkova H, Hlubocka Z, Praveckova A, Polednova A, Sukupova L, Blaha M, Maly J, Honsova E, Sedmera D, Penicka M. New Imaging Markers of Clinical Outcome in Asymptomatic Patients with Severe Aortic Regurgitation. J Clin Med. 2019 Oct 11;8(10):1654. doi: 10.3390/jcm8101654. PMID 31614523
- [Result] Steeds RP, Myerson SG. Imaging assessment of mitral and aortic regurgitation: current state of the art. Heart. 2020 Nov;106(22):1769-1776. doi: 10.1136/heartjnl-2019-316216. Epub 2020 Aug 17. No abstract available. PMID 32817242
- [Result] Kockova R, Kacer P, Pirk J, Maly J, Sukupova L, Sikula V, Kotrc M, Barciakova L, Honsova E, Maly M, Kautzner J, Sedmera D, Penicka M. Native T1 Relaxation Time and Extracellular Volume Fraction as Accurate Markers of Diffuse Myocardial Fibrosis in Heart Valve Disease - Comparison With Targeted Left Ventricular Myocardial Biopsy. Circ J. 2016 Apr 25;80(5):1202-9. doi: 10.1253/circj.CJ-15-1309. Epub 2016 Mar 17. PMID 26984717
- [Result] Zoghbi WA, Adams D, Bonow RO, Enriquez-Sarano M, Foster E, Grayburn PA, Hahn RT, Han Y, Hung J, Lang RM, Little SH, Shah DJ, Shernan S, Thavendiranathan P, Thomas JD, Weissman NJ. Recommendations for Noninvasive Evaluation of Native Valvular Regurgitation: A Report from the American Society of Echocardiography Developed in Collaboration with the Society for Cardiovascular Magnetic Resonance. J Am Soc Echocardiogr. 2017 Apr;30(4):303-371. doi: 10.1016/j.echo.2017.01.007. Epub 2017 Mar 14. No abstract available. PMID 28314623
- [Result] Vecera J, Bartunek J, Vanderheyden M, Kotrc M, Kockova R, Penicka M. Three-dimensional echocardiography-derived vena contracta area at rest and its increase during exercise predicts clinical outcome in mild-moderate functional mitral regurgitation. Circ J. 2014;78(11):2741-9. doi: 10.1253/circj.cj-14-0183. Epub 2014 Oct 3. PMID 25283687